CLINICAL TRIAL: NCT03361761
Title: Impact of a Therapeutic Education Program Specifically Adapted to the Precarious People Supported in Therapeutic Coordination Apartments on the Acceptance of Their Disease and the Management of Their Care
Brief Title: Impact of a Therapeutic Education Program on the Acceptance of Disease and Management of Care
Acronym: EDUPACT
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0108
Record Dates: First submitted 2017-11-20; First posted 2017-12-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Disease
Keywords: Chronic disease; precariousness and vulnerability; Health education
MeSH Terms: conditions — Chronic Disease; Health Education

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental: therapeutic coordination apartments with formalized/official Health education program
  Interventions: Other: Health education program
- active comparator: therapeutic coordination apartments without formalized/official Health education program
  Interventions: Other: Health education program

INTERVENTIONS:
Other: Health education program — formalized/official Health education program
  Groups: experimental
Other: Health education program — non formalized/official Health education program
  Groups: active comparator

SUMMARY:
Through its patient-centered approach and focus on developing coping skills and coping strategies, Health Education could be an effective approach in therapeutic coordination apartments to reduce the perceived treatment burden among people in precarious situations with one or more chronic diseases. Decreasing perception of burden would improve their quality of life and adherence to treatment.

The general hypothesis explored in this project is that the experience of the disease, the perception of the burden of treatment, the autonomy and the quality of life of the residents improve more importantly in therapeutic coordination apartments having implemented a formalized and structured Health Education approach (experimental group) than in those who did not set up formalized and structured Health Education approach (control group).

DETAILED DESCRIPTION:
Context: The significant increase in the number of patients with chronic disease in France in recent years has led to the implementation of therapeutic patient education programs to develop their independence and quality of life in regard to their illness. Despite this growth, socio-economic status, cultural level or education still remain significant obstacles to access to Health education for patients with psychosocial vulnerability. In this context, the implementation of an Health education approach in specific living devices called therapeutic coordination apartments (TCA) was tested in 2011. The TCAs are medico-social establishments offering accommodation and temporary medical-psycho-social support to people in a situation of precariousness affected by at least one disabling chronic pathology in order to restore their autonomy. However, only two TCAs currently offer Health Education programs integrated with their activities. These two structures were supported by the Transverse Unit for Therapeutic Education (UTET) of the University Hospital of Nantes for the construction of these programs, now authorized by the Regional Health Agency of the Pays de la Loire and effective for 18 months.

Objective: The overall objective of the project is to evaluate the added value of integrated Health Education in TCA care. The main objective will be to compare, at 6 months of care, the perception of the burden of treatment among TCA residents integrating the practice of Health Education versus control group TCA residents. The burden of treatment is defined as the perception of the constraints on daily life related to all of what a person does to heal. The secondary objectives will be, on the one hand, to evaluate the impact of Health Education in TCA on: the state of health of the residents and the perception of their state of health, their quality of life and their empowerment. On the other hand, they will study the benefits, the brakes and the levers perceived by the teams that have integrated the Health Education in their activity.

METHOD: This is a pragmatic, controlled, quasi-experimental intervention trial comparing two groups of residents: one experimental group in two TCAs incorporating Health Education and one group of 4 control TCAs. The study will be mixed, qualitative and quantitative with residents and professionals. All new volunteer residents entering TCA for 1 year will be solicited (approximately 5 to 15 per TCA). The burden of treatment will be assessed for each group after 1 month in TCA (baseline) and then at 6 months by the Treatment Burden Questionnaire. The secondary criteria will be explored quantitatively at 1 month, 6 months and 12-18 months by the EQ-5D questionnaire, the 2 global items of the WHO-QOL Brief and the MAP13, as well as the count of hospitalizations and Resident emergencies, in relation to their chronic pathology. A qualitative survey consisting of individual interviews with residents and focus groups with Therapeutic Coordination Apartments' teams practicing Health Education. The total duration of the study is 36 months.

Perspectives: By showing a potential added value for the residents of the integration of Health Education within the TCAs, this project will confirm the interest to cross specific practices of care in TCA (adapted to the precarious people, having a low level of health literacy) with Health Education practices tailored to people with multiple pathologies. The study of the perceptions of teams integrating Health Education into their practice may encourage the diffusion of these still rare programs in these structures.

ELIGIBILITY:
Inclusion Criteria:

- residents admitted in therapeutic coordination apartments since October 2017;

* with one or more chronic disease
* over 18
* accepting being enrolled in the study

Exclusion Criteria:

* residents in situation of great psychological and / or physical suffering
* Residents with diseases incompatible with questionnaires (cognitive disorders, impaired comprehension or severe speech disorder)
* Residents non-francophone without interpreter
* Residents under justice protective measure
* Investigator declining the participation of a resident for any substantial reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focuses on patients in a precarious situation with chronic pathology (one or more) that are admitted in a Therapeutic Coordination Apartment (TCA). TCA's residents are women or men, French or coming from abroad, needing medical-social welfare support to manage their disease, treatments, everyday life, and approaches.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
evaluation of the impact of a formal approach to therapeutic patient education on the intensity of the treatment burden perceived by residents compared to therapeutic coordination apartment residents not benefiting from an authorized program | 6 months after the enrolment in the study
  The Baseline assessment and the 6 months assessment of Treatment burden score (assessed with TBQ:Treatment burden survey)

SECONDARY OUTCOMES:
impact of therapeutic patient education on residents' level of depression | 6 months after the enrolment in the study
  comparison between assessments at baseline and after 6 months - (self-assessed by residents with Hospital Anxiety and Depression scale :HAD scale)
impact of therapeutic patient education on residents' health status | 6 months after the enrolment in the study
  comparison between assessments at baseline and after 6 months - (assessed with number of admission in emergency unit, number of hospitalizations)
impact of therapeutic patient education on residents' empowerment level | 6 months after the enrolment in the study
  comparison between assessments at baseline and after 6 months - (self-assessed by residents with Patient Actvation Measure survey (MAP13))
impact of therapeutic patient education on residents' perception of health status | 6 months after the enrolment in the study
  comparison between assessments at baseline and after 6 months - (self-assessed by residents with The World Healyh Organisation Quality of Life survey (WHO-QoL))
impact of therapeutic patient education on residents' quality of life | 6 months after the enrolment in the study
  comparison between assessments at baseline and after 6 months - (self-assessed by residents with Euroqol 5 dimensions survey (EQ-5D))

CONTACTS AND LOCATIONS:
Overall Officials: Clément Le Glatin, PH, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - Act Passerelle, La Roche-sur-Yon
  - Act Acothe, Le Mans
  - Act Aurore, Nantes
  - CHU de Nantes, Nantes
  - ACT Le Logis Montjoie, Nantes
  - ACT Louis Guilloux, Rennes